CLINICAL TRIAL: NCT02315599
Title: Follow-Up Evaluation for Gene-Therapy Related Delayed Adverse Events After Participation in Pediatric Oncology Branch Clinical Trials
Brief Title: Follow-Up Evaluation for Gene-Therapy-Related Delayed Adverse Events After Participation in Pediatric Oncology Branch Clinical Trials
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150028; 15-C-0028
Record Dates: First submitted 2014-12-11; First posted 2014-12-12 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01-09

CONDITIONS: Pediatric Cancers; Hematologic Malignancies; Solid Tumors
Keywords: Replication Competent Retrovirus (RCR); Replication Competent Lentivirus (RCL); T Cell Persistence; Natural History
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients screening for, participating in, or have participated in a POB gene therapy clinical trial and have received/or be scheduled to receive a genetically engineered cellular therapy.
  Interventions: Drug: anti-CD19 CAR

INTERVENTIONS:
Drug: anti-CD19 CAR

SUMMARY:
Background:

- Gene therapy involves changing the genes inside the body s cells to stop disease. It is very closely regulated. People who have had this therapy may have problems months or even years later. Researchers do not know the long-term side effects, so they want to study people who have had the therapy. They want the study to continue over the next 15 years.

Objective:

- To study over time the negative side effects from genetically engineered cellular therapy. This will be studied in people who have been in Pediatric Oncology Branch (POB) gene therapy trials.

Eligibility:

- People who are currently or were previously in a research study with gene therapy in the National Cancer Institute POB.

Design:

* Participants blood will be tested right before they get the genetically changed cells. They will get the cells as part of another study.
* For the next year, they will come back to the clinic or see their doctor at home at least every 3 months. They will answer questions about their health and blood will be drawn.
* For the next 5 years, they will go to the clinic or see their own doctor once a year. They will have physical exam and blood will be drawn.
* For 10 years after that, they will be asked every year for health information.
* Participants will keep their contact information up to date with researchers. They may be phoned for more health information.
* If the participant was under 18 years old when given the gene therapy and turns 18 during this follow-up, they will be asked to sign a new consent form when they turn 18.

DETAILED DESCRIPTION:
Background:

* Study subjects exposed to gene therapy interventions may be at risk for delayed or longterm adverse consequences. The U.S. Food and Drug Administration (FDA) has issued Long Term Follow-up After Administration of Human Gene Therapy Products: Guidance for Industry and Testing of Retroviral Vector-Based Human Gene Therapy Products for Replication Competent Retrovirus During Product Manufacture and Patient Follow-up: Guidance for Industry, which outlines a framework to assess the risk of gene therapy-related delayed adverse events and the essential elements appropriate for the conduct of long-term follow up observations.
* Accordingly, some vector designs (i.e. use of an adenovirus), based on duration of persistence accompanied by cumulative preclinical and clinical evidence, may require shorter periods of observation than other vector designs (i.e. use of a lentivirus).

Objective:

-To conduct long term safety evaluations for adverse events associated with genetically engineered cellular therapy in subjects who have participated in Pediatric Oncology Branch (POB) clinical trials.

Eligibility:

-Subjects who are planned to receive or have received at least one dose of a genetically engineered cellular therapy on a POB gene therapy clinical trial are eligible to participate.

Design:

* Subjects will be evaluated for long term safety and occurrence of adverse events according to the requirements established by the FDA guidance and the NIH Guidelines for Research Involving Recombinant or Synthetic Nucleic Acid Molecules (NIH Guidelines), to include:
* Long term follow-up after genetically engineered cellular therapy may include:

  * Post-cell infusion evaluations for T-Cell persistence (if applicable)
  * Monitoring for replication-competent retrovirus (RCR) or replication-competent lentivirus (RCL)
  * Physical examination
  * Questionnaire to detect delayed adverse events
  * Medical record review related to long term adverse events
* To ensure adequate follow up for participants in POB receiving genetically engineered cellular therapy, a maximum accrual of 500 participants will be allowed on this study. To accommodate up to 15-year follow-up of participants, this study will remain open until 2050.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must be identified eligible for, participating in, or have participated in a POB genetically engineered cellular therapy clinical trial and have received/or be scheduled to receive a genetically engineered cellular therapy.
* All monitoring and testing described in this protocol will pertain ONLY to genetically engineered cellular therapy received at the National Institutes of Health (NIH). RCR/RCL monitoring and persistence will NOT be followed for cells administered at another institution.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants screening for, participating in, or have participated in a POB gene therapy clinical trial and have received/or be scheduled to receive a genetically engineered cellular therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-12-23 (Actual); Primary Completion 2035-04-01 (Estimated); Study Completion 2050-08-01 (Estimated)

PRIMARY OUTCOMES:
Conduct long term safety evaluations after gene therapy | Every 3 months X 1 year then annually X 15 years
  PCR results (for RCR/RCL, gene transduced cells)

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-C-0028.html